CLINICAL TRIAL: NCT00269646
Title: Effect of a Low-Carbohydrate and High-Carbohydrate, High-Fiber Diet on Insulin Sensitivity and Risk Markers for Cardiovascular Disease in Men and Women With the Metabolic Syndrome
Brief Title: Comparison of Two Different Diets on Health Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Glenn Gaesser/Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HIC11487
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Metabolic Syndrome X
Keywords: Diet; Low-carbohydrate; Insulin; Dietary fiber; Diabetes; Cardiovascular disease
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Diabetes Mellitus; Cardiovascular Diseases | interventions — Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Low-carbohydrate and high-carbohydrate diets — Each subject will consume two different ad libitum diets, each for four weeks, with a 4-week washout period inbetween each diet.

SUMMARY:
The purpose of this study is to compare the effects of a low-carbohydrate diet and a high-carbohydrate, high-fiber diet, on insulin sensitivity and blood chemicals considered risk markers for heart disease, in persons with the metabolic syndrome.

Our primary hypothesis is that the ad libitum high-carbohydrate, high-fiber diet will significantly improve insulin sensitivity, whereas the ad libitum low-carbohydrate, low-fiber diet will not.

DETAILED DESCRIPTION:
Low-carbohydrate eating is becoming perceived as more than just a weight loss diet, but rather a means to improve health. Several studies have been published suggesting that low-carbohydrate diets may be preferable to low-fat diets for weight loss and in terms of some health markers. On the other hand, considerable evidence suggests that low-carbohydrate diets, high in fat, are associated with a number of adverse health outcomes. The health benefits of high-carbohydrate, high-fiber diets have also been demonstrated. This study is designed to assess the differences between the two different dietary strategies in terms of a number of health outcomes. Participants will consume, in random order, a non-calorie-restricted low-carbohydrate and a non-calorie-restricted high-carbohydrate, high-fiber diet for one month, with a 4-6 week washout period in between.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must meet the criteria of the metabolic syndrome, which is defined as having three or more of the following:

* Waist circumference: >94 cm for males; >80 cm for females
* Blood Pressure: >130/85 mmHg
* HDL-Chol (mg/dl): <50 women; <40 men)
* Triglycerides (mg/dl): >150
* Glucose (mg/dl): >100 2. Subjects must meet age requirement 3. Subjects must be nonsmokers 4. Subjects must be willing to provide written consent 5. Subjects must be willing to pick-up up meals at the GCRC and return uneaten food 6. Have no food allergies 7. Subjects must not be currently following any particular diet, and must not have intentionally lost weight by dieting during the previous 3 months 8. Subjects must not be taking nutritional supplements other than a daily multivitamin 9. Subjects must be willing to maintain current physical activity routine, which cannot exceed the equivalent of > 30 minutes per day of moderate-intensity activity 10. Blood hematocrit must be at least 40 for men and 36 for women.

Exclusion Criteria:

1. Does not meet the criteria for the metabolic syndrome 2. Does not meet age requirement 3. Smoker 4. Pregnancy 5. Food allergies 6. Unwillingness to provide written consent 7. Personal history of cardiovascular disease, including prior myocardial infarction, angioplasty, or bypass surgery 8. Known cardiovascular or metabolic diseases (e.g., diabetes) 9. Currently using medications to control blood pressure, lipids, or glucose 10. Currently on a diet or has attempted weight loss by dieting during the past 3 months 11. Currently taking nutritional supplements other than a daily multivitamin 12. Currently exercising more than the equivalent of 30 minutes/day of moderate-intensity physical activity 13. Currently on oral contraceptives 14. Hematocrit below 40 for men or below 36 for women 15. Baseline systolic blood pressure below 100 mmHg

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2004-11; Primary Completion 2008-02 (Actual); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity | before and after one month on each diet

SECONDARY OUTCOMES:
Total and LDL-cholesterol | before and after one month on each diet
C-reactive protein | before and after one month on each diet
Homocysteine | before and after one month on each diet
Fibrinogen | before and after one month on each diet
Cytokines IL-1, IL-2, IL-6 and TNF-alpha | before and after one month on each diet
Leukocyte adhesion molecules | before and after one month on each diet
Flow-mediated dilation | before and after one month on each diet

CONTACTS AND LOCATIONS:
Overall Officials: Glenn A Gaesser, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia General Clinical Research Center, Charlottesville, Virginia, United States